CLINICAL TRIAL: NCT04664283
Title: Drug-coated Balloon Versus Drug-eluting Stent for de Novo Lesions in Large Coronary Arteries Guided by Optical Coherence Tomography：a Prospective Multi-center Randomized Controlled Trial
Brief Title: Drug-coated Balloon Versus Drug-eluting Stent for de Novo Lesions in Large Coronary Arteries Guided by Optical Coherence Tomography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liu Bin (Other)
Responsible Party: Sponsor-Investigator, Liu Bin, Director of cardiology department., Second Hospital of Jilin University
Organization: Second Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: second hospital of Jilin U
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Angioplasty; Coronary Artery Disease
Keywords: coronary heart disease; large coronary vessel; optical coherence tomography; Drug-coated Balloon; Drug-eluting Stent
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DCB group by OCT guided (Experimental)
  Interventions: Device: DCB for de Novo Lesions in Large Coronary Arteries Guided by Optical Coherence Tomography
- DES group by OCT guided (Active Comparator)
  Interventions: Device: DCB for de Novo Lesions in Large Coronary Arteries Guided by Optical Coherence Tomography

INTERVENTIONS:
Device: DCB for de Novo Lesions in Large Coronary Arteries Guided by Optical Coherence Tomography — DCB for de Novo Lesions in Large Coronary Arteries Guided by both angiogram and Optical Coherence Tomography
  Other Names: DES for de Novo Lesions in Large Coronary Arteries Guided by Optical Coherence Tomography

SUMMARY:
OCT allows precise evaluation of intimal injury after lesion preparation and may improve the acute results and long-term outcomes after paclitaxel drug-coated balloon angioplasty. This prospective multicenter randomized controlled study aims to evaluate the long-term efficacy and safety of paclitaxel coated balloon in the treatment of native large coronary arteries by OCT guided is not inferior to drug-eluting stent.

ELIGIBILITY:
Inclusion Criteria:

18 to 75 years old Patients have ischemic symptoms or evidence of myocardial ischemia (inducible or spontaneous) in the presence of a stenosis of at least 50% in a native coronary artery, including stable angina, unstable angina, silent ischemia or myocardial infarction（≥1month） .

Reference vessel diameter ≥3.0 mm, and <4.5mm. Lesion length of ≤20 mm Written informed consent

Exclusion Criteria:

Myocardial infarction within 4 weeks, including ST-elevation myocardial infarction and non-ST-elevation myocardial infarction Cardiogenic shock (systolic arterial pressure <90mmHg), congestive heart failure (NYHA=4，EF≤35%) Severe valvular heart disease Life expectancy no more than 1 year or factors causing difficulties in clinical follow up Intolerance to aspirin and/or clopidogrel, ticagrelor Known intolerance or allergy to heparin, contrast agents, paclitaxel, iopromide, rapamycin, polylactic acid-glycolic acid copolymer, Co-Cr alloy or platinum-chromium alloy Leukopenia or thrombopenia A history of peptic ulcer or GI bleeding in the previously Stroke within 6 months prior to the operation A history of severe hepatic or renal failure Stents covering a major side branch (≥2.5 mm need to intervention) Left main lesion Graft lesion Aortic-coronary ostial lesion In-stent restenotic lesion Chronic total occlusion Severe calcified lesions. Visible angiographic thrombus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
late lumen loss （LLL） | Follow-up coronary angiography at 12 months after the procedure
  late lumen loss between DCB treated group and DES treated group evaluated by quantitative coronary analysis in patients with CHD

SECONDARY OUTCOMES:
The incidence rate of device-related ischemic events | Clinical follow up at 30 days, 3，6, 9 and 12 months after the procedure
  The incidence rate of device-related ischemic events including cardiovascular death, target vessel related myocardial infarction and ischemia-driven revascularization between DCB treated group and DES treated group
The incidence rate of patient-related ischemic events | Clinical follow up at 30 days, 3，6, 9 and 12 months after the procedure
  TThe incidence rate of patient-related ischemic events including all myocardial infarction , any revascularization and all-cause death between DCB treated group and DES treated group

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Hospital of Jilin University, Changchun, Jilin
  - the Second hospital of Jilin University, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu Y, Zhang YJ, Deng LX, Yin ZY, Hu T, Wang Q, Li Y, Li JY, Guo WY, Mou FJ, Tao L. 12-Month clinical results of drug-coated balloons for de novo coronary lesion in vessels exceeding 3.0 mm. Int J Cardiovasc Imaging. 2019 Apr;35(4):579-586. doi: 10.1007/s10554-018-1505-z. Epub 2019 Mar 30. PMID 30929102
- [Result] Cuculi F, Young M, Beeler R, Schoenenberger AW, Erne P. Good efficacy of drug-eluting balloons in a mixed population of patients with coronary artery disease. J Invasive Cardiol. 2012 Apr;24(4):151-3. PMID 22477748
- [Result] Lu W, Zhu Y, Han Z, Sun G, Qin X, Wang Z, Liu G, Xi W, Wang X, Pan L, Qiu C. Short-term outcomes from drug-coated balloon for coronary de novo lesions in large vessels. J Cardiol. 2019 Feb;73(2):151-155. doi: 10.1016/j.jjcc.2018.07.008. Epub 2018 Oct 23. PMID 30366637
- [Result] Yu X, Ji F, Xu F, Zhang W, Wang X, Lu D, Yang C, Wang F. Treatment of large de novo coronary lesions with paclitaxel-coated balloon only: results from a Chinese institute. Clin Res Cardiol. 2019 Mar;108(3):234-243. doi: 10.1007/s00392-018-1346-8. Epub 2018 Aug 3. PMID 30074078
- [Result] Lansky A, Wijns W, Xu B, Kelbaek H, van Royen N, Zheng M, Morel MA, Knaapen P, Slagboom T, Johnson TW, Vlachojannis G, Arkenbout KE, Holmvang L, Janssens L, Ochala A, Brugaletta S, Naber CK, Anderson R, Rittger H, Berti S, Barbato E, Toth GG, Maillard L, Valina C, Buszman P, Thiele H, Schachinger V, Baumbach A; TARGET All Comers Investigators. Targeted therapy with a localised abluminal groove, low-dose sirolimus-eluting, biodegradable polymer coronary stent (TARGET All Comers): a multicentre, open-label, randomised non-inferiority trial. Lancet. 2018 Sep 29;392(10153):1117-1126. doi: 10.1016/S0140-6736(18)31649-0. Epub 2018 Sep 3. PMID 30190206
- [Result] Cortese B, Silva Orrego P, Agostoni P, Buccheri D, Piraino D, Andolina G, Seregni RG. Effect of Drug-Coated Balloons in Native Coronary Artery Disease Left With a Dissection. JACC Cardiovasc Interv. 2015 Dec 28;8(15):2003-2009. doi: 10.1016/j.jcin.2015.08.029. Epub 2015 Nov 25. PMID 26627997
- [Result] Nishiyama N, Komatsu T, Kuroyanagi T, Fujikake A, Komatsu S, Nakamura H, Yamada K, Nakahara S, Kobayashi S, Taguchi I. Clinical value of drug-coated balloon angioplasty for de novo lesions in patients with coronary artery disease. Int J Cardiol. 2016 Nov 1;222:113-118. doi: 10.1016/j.ijcard.2016.07.156. Epub 2016 Jul 27. PMID 27494722